CLINICAL TRIAL: NCT04586699
Title: Meditation Accelerated Brain Stimulation for Depression
Acronym: MediTMS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jyoti Mishra, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MediTMS
Record Dates: First submitted 2020-09-30; First posted 2020-10-14 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Medi1TMS (Experimental): rTMS theta-burst protocol paired with a consistent attention-to-breath task
  Interventions: Device: Medi1TMS
- Medi2TMS (Active Comparator): rTMS theta-burst protocol paired with an intermittent deep breathing task
  Interventions: Device: Medi2TMS

INTERVENTIONS:
Device: Medi1TMS — rTMS theta-burst protocol paired with a consistent attention-to-breath task
  Arms: Medi1TMS
Device: Medi2TMS — rTMS theta-burst protocol paired with an intermittent deep breathing task
  Arms: Medi2TMS

SUMMARY:
Repetitive Transcranial magnetic stimulation (rTMS) is an FDA-approved treatment for depression that involves brief magnetic stimulation pulses on the dorsolateral prefrontal cortex (DLPFC) brain region. The ultimate goal of this treatment is to increase excitability and long-term plasticity in DLPFC, a brain region shown to be hypo-active in depression. Unfortunately, rTMS only has low to moderate efficacy; remission rates for patients range from ~15-30% in large randomized controlled trials. The focus of this research is to develop a next-generation rTMS protocol that is guided by the basic principles underlying brain plasticity, in order to improve the efficacy of rTMS for the treatment of depression. Specifically, in this study the investigators will test rTMS paired with a depression-relevant cognitive state of internal attention.

DETAILED DESCRIPTION:
Repetitive Transcranial magnetic stimulation (rTMS) is an FDA-approved treatment for depression that involves brief magnetic stimulation pulses on the dorsolateral prefrontal cortex (DLPFC) brain region. The ultimate goal of this treatment is to increase excitability and long-term plasticity in DLPFC, a brain region shown to be hypo-active in depression. Unfortunately, rTMS only has low to moderate efficacy; remission rates for patients range from ~15-30% in large randomized controlled trials. The focus of this research is to develop a next-generation rTMS protocol that is guided by the basic principles underlying brain plasticity, in order to improve the efficacy of rTMS for the treatment of depression. Specifically, in this study the investigators will test rTMS paired with a depression-relevant cognitive state of internal attention. Meditative internal focus has been shown to benefit depression. Our own research shows that the neural correlates of attention-to-breath are associated with greater mindfulness. Hence, in this study we will pair breath training with rTMS neuro-stimulation.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe depression (PHQ-9 scale score >9 with confirmation using the Structured Clinical Interview for DSM-5 Disorders)
* treatment refractory to antidepressants (i.e. failed 1-3 antidepressants in current episode) or intolerant to antidepressants (i.e. tried 2 antidepressant of inadequate dose/duration in current episode)

Exclusion Criteria:

* active substance abuse/dependence
* psychotic disorders
* any factor that increases risk of TMS (metal implants/history of stroke/seizure disorder).
* displaying acutely suicidal behaviors on the Columbia Suicide Severity Rating Scale.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Clinical Depression (Remission) | up to 6 weeks
  PHQ9 depression scale
Change from baseline brain activity in attention-to-breath task | up to 6 weeks
  Electroencephalography (EEG) power in attention-to-breath task

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti Mishra, PhD, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - Neuromodulation Clinic Veterans Affairs San Diego, San Diego, California
  - UC San Diego Health Psychiatry, San Diego, California

IPD SHARING:
Plan to Share IPD: Yes
De-identified raw and processed data will be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: At time of publication
Access Criteria: The PI will review sharing requests and provide access to researchers.

DOCUMENTS (1):
  • Informed Consent Form (2025-01-26): https://cdn.clinicaltrials.gov/large-docs/99/NCT04586699/ICF_000.pdf